CLINICAL TRIAL: NCT04408118
Title: Phase II Clinical Trial to Evaluate the Efficacy and Safety of First Line Atezolizumab in Combination With Paclitaxel and Bevacizumab (Avastin®) in Patients With Advanced or Metastatic Triple-negative Breast Cancer
Brief Title: First Line Atezolizumab, Paclitaxel, and Bevacizumab (Avastin®) in mTNBC
Acronym: ATRACTIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP150; 2019-001503-20 (EudraCT Number)
Record Dates: First submitted 2020-05-20; First posted 2020-05-29 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer; Triple Negative Breast Cancer
Keywords: breast cancer; metastatic breast cancer; triple negative breast cancer; HER2 negative; HR negative
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — atezolizumab; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Paclitaxel + Bevacizumab (Avastin®) (Experimental): All eligible patients will be treated with atezolizumab (840 mg) intravenously on days 1 and 15, Paclitaxel (90 mg/m2) on days 1, 8 and 15 via IV infusion and Bevacizumab (Avastin® 10mg/kg) intravenously on days 1 and 15.
  Treatment cycles and patient visits are organized in scheduled cycles of 28 days.
  Interventions: Drug: Atezolizumab; Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab (840 mg) will be administered intravenously on Days 1 and 15.
  The first infusion of atezolizumab will be administered over 60 minutes. If the first infusion is tolerated, all subsequent infusions may be delivered over 30 minutes.
Drug: Paclitaxel — Will be administered on days 1, 8 and 15 via IV infusion over 1 hour.
Drug: Bevacizumab — Will be administered intravenously over 30-90 minutes on Days 1 and 15.
  Other Names: Avastin

SUMMARY:
This is a multicenter, open-label, single-arm, phase II clinical trial to evaluate to evaluate the efficacy and safety of first line atezolizumab in combination with paclitaxel and bevacizumab (Avastin®) in patients with advanced or metastatic triple-negative breast cancer (mTNBC)

DETAILED DESCRIPTION:
Men and women age ≥ 18 years with previously untreated unresectable locally advanced or metastatic triple-negative breast cancer (TNBC) that is not amenable to resection with curative intent regardless of programmed death-ligand 1 (PD-L1) status.

The number of patients to be included is 100 patients. The primary objective is to evaluate the efficacy -in terms of progression-free survival (PFS)- of first line atezolizumab in combination with paclitaxel and bevacizumab (Avastin®) in patients with unresectable locally advanced or metastatic TNBC.

After signing the ICF and confirmed eligibility, patients will begin treatment on 28 days cycles: Atezolizumab (840 mg) intravenously on days 1 and 15; Paclitaxel (90 mg/m2) via IV infusion on days 1, 8 and 15; Bevacizumab (Avastin® 10mg/kg) intravenously on days 1 and 15.

Patients will receive treatment until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

Patients discontinuing the study treatment will enter a post- treatment follow-up period until death, withdrawal of consent, patient is lost to follow-up, or study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) prior to participation in any study-related activities.
2. Male or female patients ≥ 18 years at the time of signing ICF.
3. Ability to comply with the study protocol, in the investigator's judgment.
4. Histologically confirmed TNBC -regardless of PD-L1 status- per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) criteria based on local testing on the most recent analyzed biopsy. Triple-negative is defined as <1% expression for estrogen receptor (ER) and progesterone receptor (PgR) as determined by immunohistochemistry (IHC), and negative for HER2 (0-1+ by immunohistochemistry [IHC] or 2+ and negative by in situ hybridization [ISH] test).
5. Unresectable locally advanced or metastatic disease documented by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to resection with curative intent.
6. No prior chemotherapy and/or targeted therapy and/or immunotherapy and/or antiangiogenic agent for triple negative MBC. Patients who have received (neo)adjuvant taxane-based chemotherapy and/or immunotherapy and/or an antiangiogenic agent are required to have a disease-free interval (DFI) of at least 12 months after completion of each of these treatments. For (neo)adjuvant non-taxane-based chemotherapy, a DFI of at least 6 months is required.
7. Resolution of all acute toxic effects of prior anti-cancer therapy to grade ≤ 1 as determined by the NCI-CTCAE v.5.0 (except for alopecia, grade ≤ 2 peripheral neuropathy, or other toxicities not considered a safety risk for the patient at investigator's discretion).
8. Evidence of measurable disease or non-measurable disease as per RECIST v.1.1. Patients with only bone lesions are also eligible.
9. Willingness and ability to provide the most recent tumor biopsy since last progression from either metastatic or primary tissues at the time of the inclusion to perform exploratory studies. If not feasible, patient eligibility should be evaluated by a Sponsor's qualified designee. An additional tumor biopsy from either metastatic or primary (only if metastatic biopsies cannot be obtained for inaccessible lesion or subject safety concern) tissues will be collected as soon as possible at disease progression or study termination whenever it is feasible.

   Note: Patients for whom tumor biopsies cannot be obtained (e.g., inaccessible tumor or safety concern) may submit archived pathological material from either metastatic or primary sites, but the most recent tumor biopsy from the patient should be obtained when available.

   Note 2: Bone biopsies are only acceptable if performed on bone metastases with associated soft tissue mass, where the biopsy is performed on the soft tissue mass, and a decalcification process is not used. Cytology samples and decalcified bone specimens are unacceptable due to lack of validation studies.
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
11. Life expectancy of ≥12 weeks.
12. Adequate hematologic and organ function within 14 days before the first study treatment on Cycle 1 Day 1 (C1D1), defined by the following parameters:

    a. Hematological: i. White blood cell (WBC) count > 3.0 x 109/L. ii. Absolute neutrophil count (ANC) > 1.5 X 109/L (without granulocyte colony-stimulating factor [G-CSF] support within 2 weeks prior to Cycle 1 Day1) iii. Lymphocyte count ≥ 0.5 x 109/L (500 cells/uL) iv. Platelet count ≥ 75.0 x 109/L (without transfusion within 2 weeks prior to Cycle 1 Day 1) v. Hemoglobin > 9.0 g/dL (Patients may be transfused or receive erythropoietic treatment to meet this criterion).

    Note: Patients cannot be transfused platelets within 14 days prior to C1D1 to meet this criterion. The use of G-CSF within 14 days prior to C1D1 is also prohibited.

    b. Hepatic: Total bilirubin ≤ 1.5 times the upper limit of normal (× ULN) (≤ 3 x ULN in the case of Gilbert's disease); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN (in the case of liver metastases ≤ 5 × ULN); alkaline phosphatase (ALP) ≤ 2.5 × ULN (≤ 5 × ULN in the case of liver and/or bone metastases).

    c. Serum albumin ≥ 2.5 g/dL

    d. Renal: Serum creatinine < 1.5 × ULN or creatinine clearance ≥ 50 mL/min based on Cockcroft-Gault glomerular filtration rate estimation. No proteinuria by urinalysis. In cases of proteinuria > ULN by urinalysis, proteinuria should be less than 500 mg by 24-hour urine collection.

    e. Coagulation:
    * For patients not receiving therapeutic anticoagulation: Partial Thromboplastin Time (PTT) (or activated Partial Thromboplastin Time [aPTT]) and International Normalized Ratio (INR) ≤ 1.5 × ULN.
    * For patients receiving therapeutic anticoagulation: Stable anticoagulant regimen.
13. Negative human immunodeficiency virus (HIV) test at screening. Patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200 cells/uL, and have an undetectable viral load.
14. Negative hepatitis B surface antigen (HBsAg) test and negative total hepatitis B core antibody (HBcAb) tests at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. Current treatment with anti-viral therapy for HBV is not allowed.

    Note: HBV DNA test only to be performed for patients with a positive total HBcAb test.
15. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening.

    Note: HCV RNA test only to be performed for patients with a positive HCV antibody test.
16. Women of childbearing potential must have a negative serum pregnancy test within 14 days before study treatment initiation and agree to remain abstinent (refrain from heterosexual intercourse) or use one highly effective contraceptive method, or two effective contraceptive methods, for at least 5 months after the last dose of atezolizumab, and for at least 6 months after the last dose of paclitaxel and bevacizumab, whichever is later.

Men with female partners of childbearing potential or pregnant female partners, must remain abstinent or use a condom during the treatment period and for at least 5 months after the last dose of atezolizumab, and for at least 6 months after the last dose of paclitaxel and bevacizumab, whichever is later, to avoid exposing the embryo. Men must refrain from donating sperm during this same period. Due to the possibility of irreversible infertility with paclitaxel, men receiving this chemotherapy should consult with their doctor regarding conservation of sperm prior to treatment initiation.

Exclusion Criteria:

1. Known active uncontrolled or symptomatic central nervous system (CNS) metastases as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases are eligible if they meet the following criteria:

   * Evidence of measurable disease or non-measurable disease as per RECIST v.1.1.
   * The patient has no history of intracranial hemorrhage.
   * The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
   * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted.
2. History of leptomeningeal disease.
3. Uncontrolled tumor-related pain. Note 1: Patients requiring pain medication must be on a stable regimen at study entry.

   Note 2: Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrolment. Patients should be recovered from the effects of radiation.
4. Active or history of autoimmune disease or immune deficiency, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis for a more comprehensive list of autoimmune diseases and immune deficiencies, with the following exceptions:

   * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
   * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   * Patients with eczema, psoriasis, lichen simplex chronicum, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

     * Rash must cover < 10% of body surface area.
     * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
     * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.

   Note: Patients with indwelling catheters (e.g., PleurX® are allowed)
6. Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L; calcium >12 mg/dL).
7. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.

   Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
8. Active tuberculosis.
9. Significant cardiovascular disease 6 months prior to initiation of study treatment. These include New York Heart Association Class II or greater cardiac disease, myocardial infarction, unstable arrhythmia, or unstable angina, symptomatic pericarditis, ventricular arrhythmias (except for benign premature ventricular contractions), arrhythmias or conduction abnormalities requiring a pacemaker or not controlled with medication, and prior peripheral vascular disease including any cerebrovascular accident including transient ischemic attack, any pulmonary embolism, any prior deep vein thrombosis, and/or any grade ≥ 2 peripheral vascular disease.
10. Left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO).
11. Uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and diastolic blood pressure greater than 100 mmHg).
12. Major surgical procedure (defined as requiring general anesthesia) or significant traumatic injury within 28 days of start of study drug, or patients who have not recovered from the side effects of any major surgery.
13. Concurrent malignancy(ies) or malignancy(ies) within 5 years prior to study enrollment except for carcinoma in situ of the cervix, non-melanoma skin carcinoma, or stage I uterine cancer. For other cancers considered to have a low risk of recurrence, discussion with the Medical Monitor is required.
14. Treatment with therapeutic oral or intravenous (IV) antibiotics or severe infection within 2 weeks prior to initiation of study treatment.

    Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
15. Prior allogeneic stem cell or solid organ transplantation.
16. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months the final dose of atezolizumab.
17. Extracranial radiotherapy or limited-field palliative radiotherapy within seven days prior to study enrolment, or patients who have not recovered from radiotherapy-related toxicities to baseline or grade ≤ 1.
18. Treatment with investigational therapy within 28 days prior to initiation of study treatment.
19. Treatment with systemic immunosuppressive medication 2 weeks prior to initiation of study treatment (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    Note 1: Patients who have received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor approval has been obtained.

    Note 2: Patients who are receiving mineralocorticoids (e.g., fludrocortisone), inhaled corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
20. Chronic daily intake of antiplatelet drugs (e.g., aspirin doses of 325 mg/day or higher or non-steroidal anti-inflammatory medication known to inhibit platelet function).
21. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion protein.
22. Breast-feeding women.
23. Any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgement, contraindicate patient participation in the clinical study.
24. Concurrent participation in other interventional clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
PFS (Progression-free Survival) | 24 months
  From a clinical point of view, the primary endpoint for this study is the PFS (progression-free survival) defined as the period of time from treatment initiation to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined locally by the investigator using RECIST v.1.1.

SECONDARY OUTCOMES:
Efficacy (TTR) | 24 months
  TTR is defined as the time from the treatment initiation to time of the first objective tumor response (tumor shrinkage of ≥30%) observed for patients who achieved a complete response (CR) or partial response (PR).
Efficacy (ORR) | 24 months
  Objective response rate (ORR) is defined as the sum of CR and PR relative to the number of patients in the analysis set with measurable disease at baseline.
Efficacy (CBR) | 24 months
  Clinical benefit rate (CBR) is defined as the proportion of participants with CR, PR or SD ≥24 weeks relative to the number of patients in the analysis set.
Efficacy (DoR) | 24 months
  Duration of response (DoR) is defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression, death due to any cause or treatment discontinuation, whichever occurs first.
Efficacy (OS) | 24 months
  Overall survival (OS) is defined as the time from date of treatment initiation to date of death due to any cause. In the absence of confirmation of death, survival time will be censored to last date the participant was known to be alive.
Efficacy (Best percentage of change of target tumor lesions) | 24 months
  Best percentage of change from baseline in the size of target tumor lesions is defined as the biggest decrease, or smallest increase if no decrease will be observed.
Safety AEs and SAEs | 24 months
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs) according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5.0, including dose reductions, delays, and treatment discontinuations.
Exploratory objectives (irPFS) | 24 months
  Immune-related progression-free survival (irPFS) is defined as the period of time from the date of treatment initiation to the date of the first documentation of objective progression of disease (irPD) or death due to any cause in absence of documented irPD.
Exploratory objectives (irORR) | 24 months
  Immune-related objective response (irORR) is defined as the proportion of participants with irCR or irPR relative to the number of patients in the analysis set with measurable disease at baseline.
Exploratory objectives (molecular markers) | 24 months
  Changes in mutation and copy number in oncogenes, tumor suppressors, and/or other genes associated with disease progression assessed in liquid biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, PhD, Principal Investigator — MedSIR
Locations (26):
- France (3):
  - Hopital Europeen Georges Pompidou, Paris
  - Hôpital Tenon AP-HP, Paris
  - Insitut de cancérologie Strasbourg Europe, Strasbourg
- Germany (3):
  - Klinikum Dessau (MVZ) - Frauenheilkunde, Dessau
  - University Hospital Essen, Essen
  - Universitätsklinikum Mannheim, Mannheim
- Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Naples, Italy
- Spain (17):
  - Hospital de Dénia-MarinaSalud, Denia, Alicante
  - Hospital Universitario La Ribera, Alzira
  - Hospital de Sant Joan Despí - Moises Broggi, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital Ruber Juan Bravo, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson Cancer Center, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario San Juan de Alicante, Sant Joan d'Alacant
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Quirón Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Royal Cornwall Hospitals Nhs Trust, Truro

REFERENCES:
- [Derived] Gion M, Blancas I, Cortez-Castedo P, Cortes-Salgado A, Marme F, Blanch S, Morales S, Diaz N, Calvo-Plaza I, Recalde S, Martinez-Bueno A, Ruiz-Borrego M, Llabres E, Taberner MT, de Laurentiis M, Garcia-Vicente S, Guerrero JA, Boix O, Rodriguez-Morato J, Sampayo-Cordero M, Antonarelli G, Perez-Garcia JM, Cortes J, Llombart-Cussac A; ATRACTIB Trial Investigators. Atezolizumab plus paclitaxel and bevacizumab as first-line treatment of advanced triple-negative breast cancer: the ATRACTIB phase 2 trial. Nat Med. 2025 Aug;31(8):2746-2754. doi: 10.1038/s41591-025-03734-3. Epub 2025 Jun 4. PMID 40467896
- [Derived] Agostinetto E, Eiger D, Punie K, de Azambuja E. Emerging Therapeutics for Patients with Triple-Negative Breast Cancer. Curr Oncol Rep. 2021 Mar 24;23(5):57. doi: 10.1007/s11912-021-01038-6. PMID 33763756